CLINICAL TRIAL: NCT06869538
Title: Effect of Pilates and Kegel Exercises During Pregnancy on Postpartum Urinary and Fecal Incontinence and Women's Quality of Life
Brief Title: Effect of Pilates and Kegel Exercises During Pregnancy
Status: Completed | Type: Observational
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Guner CICEK, Associate Professor, Hitit University
Other Study IDs: 469; Hitit University (Other: Hitit University)
Record Dates: First submitted 2025-02-08; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy
Keywords: Urinary İncontinence; Fecal İncontiance; Quality Of Life; pregnancy; exercise
MeSH Terms: conditions — Nocturnal Enuresis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exercise — For the Pilates exercises, a Pilates instructor created movements (squeeze mini ball, stretch hoop, circle with large ball, back and forth with large ball, and squat) in the gymnasium of the pregnancy school for 8 weeks, 2 days a week. Auxiliary equipment (mini ball, resistance band, Pilates ring) was used. Kegel exercises were performed 4 days a week, 3 sessions a day for 8 weeks.

SUMMARY:
Urinary incontinence and fecal incontinence are common health problems in the postpartum period because of their effect on daily life and are likely to reduce quality of life. It is known that the most effective way to protect from UI during pregnancy and the postpartum period is pelvic floor muscle exercise. This study aimed to investigate the effects of Pilates and Kegel exercises applied during pregnancy on the quality of life of urinary and fecal incontinence in the postpartum period.

DETAILED DESCRIPTION:
In this study; the effects of pilates and kegel exercises on urinary and fecal incontinence of pregnant women in the 1st and 3rd months postpartum are investigated and which of the applied pilates and kegel exercises is more effective on urinary and fecal quality of life.67 pregnant women with a mean age of 27.29±3.27 years participated in the study. Pilates exercise group (PEG, n=24), Kegel exercise group (KEG, n=22), and Control group (CG, n=21) were formed with the purposeful method. PEG exercise programs were applied for 8 weeks, 2 days a week, 40 minutes, and KEG for 8 weeks, 4 days a week, 3 sessions per day. The groups were applied the International Incontinence Questionnaire Short Form, Urinary Incontinence Quality of Life Scale, Wexner Continence Assessment Scale, and Fecal Incontinence Quality of Life Scale at 1st. and 3rd. months postpartum

ELIGIBILITY:
Inclucision Criteria

* Being between the ages of 18-38 years,
* Not having a condition that prevents exercise,
* Being in the 3rd trimester of pregnancy,
* Voluntarily accepting to participate in the study, a
* Answering each of the scale items,
* Having a vaginal (normal) birth.

Exclusion Criteria:

* Not being between the ages of 18-38,
* Having a condition that prevents exercise,
* Not being in the 1st and 2nd trimesters of pregnancy,
* Leaving scale items blank, and having a cesarean section.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnancy women
Study Population: Pregnancy women
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2022-02-13 (Actual)

PRIMARY OUTCOMES:
Baseline Anthropometric Measurements (Weight, Height, BMI) | 2021 june
  Baseline meausurement ( 1 week) Participants will be evaluated at baseline. Data collection refers to anthropometric parameters (Weight, height and BMI. BMI BMI will calculated as weight in kilograms divided by height squared (kg/m2) in meters
Urinary Incontinence Quality of Life Scale (I-QOL)-Baseline and Follow-up Measurements | June 2021 (Baseline) and 1st and 3rd months postpartum
  Urinary Incontinence Quality of Life Scale (I-QOL) - Evaluates the quality of life related to urinary incontinence.
  Description: Evaluates the quality of life related to urinary incontinence. This scale was applied at baseline and at the 1st and 3rd months postpartum.
  Minimum Value: 0 (Poor quality of life) Maximum Value: 100 (High quality of life) Higher Scores Indicate: Better quality of life Data Aggregation: Mean ± SD and comparison of scores between groups using ANOVA.
Effect of an 8-Week Exercise Intervention on Urinary and Fecal Incontinence - Measured by ICIQ-UI Short Form and Wexner Continence Assessment Scale | Baseline (June 2021), Post-intervention (August 2021), and Follow-up at 1st and 3rd months postpartum.
  This measure evaluates the effect of an 8-week exercise intervention on urinary and fecal incontinence in pregnant women. Urinary incontinence severity will be assessed using the ICIQ-UI SF, and fecal incontinence using the Wexner Scale at baseline, post-intervention (8 weeks), and 1st and 3rd months postpartum.
  Participants are divided into two groups:
  Pilates Group (PEG): Performed Pilates twice a week, 40 minutes per session, for 8 weeks, using a mini ball, resistance band, and Pilates ring.
  Kegel Group (KEG): Performed Kegel exercises 4 days a week, 3 sessions per day, for 8 weeks, involving controlled pelvic floor contractions and relaxations.
  Measurement Tools:
  Urinary Incontinence: ICIQ-UI SF Fecal Incontinence: Wexner Scale
International Incontinence Questionnaire Short Form Score (ICIQ-SF) - Urinary Incontinence Impact | 2021 September 2021 November
  Description: Assesses the impact of urinary incontinence on daily life. Minimum Value: 0 (No impact) Maximum Value: 21 (Severe impact) Higher Scores Indicate: Worse quality of life Data Aggregation: Mean ± SD and comparison of groups using repeated measures ANOVA, paired t-test for pre- and post-intervention comparison.
Wexner Continence Assessment Scale Score - Fecal Incontinence Severity | September 2021 - November 2021
  Description: Measures the severity of fecal incontinence. Minimum Value: 0 (Complete continence) Maximum Value: 20 (Complete incontinence) Higher Scores Indicate: Worse fecal incontinence Data Aggregation: Mean ± SD and comparison of groups using repeated measures ANOVA, paired t-test for pre- and post-intervention comparison.
Fecal Incontinence Quality of Life Scale (FIQL) Score | September 2021 - November 2021
  Description: Assesses the quality of life related to fecal incontinence. Minimum Value: 1 (Poor quality of life) Maximum Value: 5 (High quality of life) Higher Scores Indicate: Better quality of life Data Aggregation: Mean ± SD and comparison of groups using repeated measures ANOVA, paired t-test for pre- and post-intervention comparison

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University, Çorum, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available
Supporting Information: Study Protocol

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29882074/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32378735/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31820378/

DOCUMENTS (1):
  • Informed Consent Form (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT06869538/ICF_000.pdf